CLINICAL TRIAL: NCT06613113
Title: A Single-arm, Single-center Clinical Study of Fruquintinib Combined With Adebrelimab and High and Low Dose Radiotherapy in the Treatment of Second-line and Above Failure MSS Metastatic Colorectal Cancer.
Brief Title: Fruquintinib Combined With Adebrelimab and High and Low Dose Radiotherapy in the Treatment of Second-line and Above Failure MSS Metastatic Colorectal Cancer.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo Medical Center Lihuili Hospital (Other Government)
Collaborators: Shanghai Shengdi Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2024PJ169
Record Dates: First submitted 2024-09-22; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-07

CONDITIONS: MSS Metastatic Colorectal Cancer
Keywords: MSS Metastatic Colorectal Cancer; Fruquintinib; Adebrelimab; High and Low Dose Radiotherapy
MeSH Terms: interventions — HMPL-013; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fruquintinib Group (Experimental): Participants will receive the combination of Fruquintinib and Adebrelimab within 3 weeks after completion of high and low dose radiotherapy on metastases until disease progression or intolerable toxicity occurred.
  Interventions: Drug: Fruquintinib

INTERVENTIONS:
Drug: Fruquintinib — After receiving high and low dose radiotherapy on metastases, the enrolled patients will receive the combination of Fruquintinib and Adebrelimab. RECIST 1.1 standard was used for clinical tumor imaging evaluation every 6 weeks (±7 days). For complete response (CR) ,partial response (PR), or stable disease (SD), the enrolled patients will continue to receive the combination of Fruquintinib and Adebrelimab. Participants will receive the combination of Fruquintinib and Adebrelimab until disease progression or intolerable toxicity occurred.
  Other Names: Adebrelimab; high and low dose radiotherapy

SUMMARY:
The goal of this clinical trial is to learn about Fruquintinib combined with Adebrelimab and high and low dose radiotherapy in the treatment of second-line and above failure MSS(microsatellite stability) metastatic colorectal cancer.

The main question it aims to answer is: The efficacy and safety of Fruquintinib combined with Adebrelimab and high and low dose radiotherapy in the third line and beyond treatment of MSS metastatic colorectal cancer.

Participants will receive the combination of Fruquintinib and Adebrelimab within 3 weeks after completion of high and low dose radiotherapy on metastases until disease progression or intolerable toxicity occurred.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, gender not limited；
2. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score 0-1；
3. Previously identified as MSS type mCRC；
4. Metastatic colorectal cancer (mCRC) with disease progression after receiving standard second-line treatment according to Chinese Society of Clinical Oncology ( CSCO) guidelines；
5. At least one measurable lesion (RECIST 1.1)；
6. Be able to adhere to the protocol during the research period；
7. Sign the informed consent form.

Exclusion Criteria:

1. For individuals with a history of uncontrolled epilepsy, central nervous system disorders, or mental disorders, the clinical severity of which may hinder the signing of informed consent forms or affect the patient's adherence to oral medication, as determined by the researcher；
2. Accompanied by other malignant tumors that have not been cured；
3. The baseline blood routine and biochemical indicators of the subject do not meet the following criteria: hemoglobin ≥ 90g/L; Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; Platelets ≥ 100 × 109/L; Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤ 2.5 times the normal upper limit; Alkaline phosphatase (ALP) ≤ 2.5 times the normal upper limit value; Serum total bilirubin<1.5 times the normal upper limit value; Serum creatinine<1 times the upper limit of normal; Serum albumin ≥ 30g/L；
4. Serious (i.e. active) heart disease in clinical practice, such as symptomatic coronary heart disease, congestive heart failure, or severe arrhythmia requiring medication intervention, or a history of myocardial infarction in the past 12 months；
5. Irreversible coagulation dysfunction or concurrent active massive bleeding；
6. Combination of active infections requiring antibiotic treatment；
7. Individuals who are allergic to any research drug ingredients；
8. Women with concurrent pregnancy or lactation；
9. Organ transplantation requires immunosuppressive therapy and long-term hormone therapy；
10. Patients with autoimmune diseases；
11. There is a history of drug treatment in previous plans。

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 1 year
  objective response rate

SECONDARY OUTCOMES:
PFS | 2 years
  Progression Free Survival
OS | 3 years
  Overall Survival
DCR | 3 years
  Disease Control Rate
DoR | 3 years
  Duration of Overall Response
AE | 3 years
  adverse event

CONTACTS AND LOCATIONS:
Locations (1):
- Kaitai Liu, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No